CLINICAL TRIAL: NCT02885519
Title: Integrated Mental Health Care and Vocational Rehabilitation to Individuals on Sick Leave Due to Burnout, Adjustment Disorder or Psychological Stress in Denmark (the Danish IBBIS Study): A Multi-center Randomized Controlled Trial
Brief Title: Integrated Mental Health Care and Vocational Rehabilitation to Individuals on Sick Leave Due to Stress Disorders
Acronym: IBBIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amager Hospital (Other)
Collaborators: The Danish Agency for Labour Market and Recruitment (Other); Copenhagen Municipality, Denmark (Other Government); Gentofte Municipality, Denmark (Unknown); Municipality of Lyngby-Taarbæk, Denmark (Unknown); Gladsaxe Municipality, Denmark (Other)
Responsible Party: Principal Investigator, Lene Falgaard Eplov, Head of Research, Associate professor, Amager Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IBBIS Stress
Record Dates: First submitted 2016-08-15; First posted 2016-08-31 (Estimated); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Adjustment Disorder; Burnout; Psychological Stress
Keywords: Vocational Rehabilitation; Common Mental Disorders; Return to Work; Mental Health Services; Psychological Stress; Adjustment Disorder; Burnout; Integration; Cognitive Behavior Therapy
MeSH Terms: conditions — Adjustment Disorders; Burnout, Psychological; Stress, Psychological | interventions — Rehabilitation, Vocational

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): Standard treatment and standard vocational rehabilitation
- IBBIS MHC (Experimental): IBBIS mental health care and standard vocational rehabilitation
  Interventions: Behavioral: IBBIS mental health care and standard vocational rehabilitation
- IBBIS integrated MCH and VR (Experimental): Integrated mental health care and vocational rehabilitation
  Interventions: Behavioral: Integrated mental health care and vocational rehabilitation

INTERVENTIONS:
Behavioral: IBBIS mental health care and standard vocational rehabilitation — Standard vocational rehabilitation.
  Stepped mental health care provided by the IBBIS mental health care team (e.g. nurses, psychologists and medical doctors) with the treatment modalities:
  Psychoeducation Bibliotherapy Stress-coaching Mindfulness-based stress reduction Monitoring and re-assessment
  Arms: IBBIS MHC
Behavioral: Integrated mental health care and vocational rehabilitation — Integrated mental health care and vocational rehabilitation provided by the IBBIS team. The IBBIS team is composed by employment specialists from the municipal job centers and health care professionals from the mental health services (e.g. nurses, psychologists, and medical doctors).
  Mental health care is provided according to a stepped care model with the following treatment modalities:
  Psychoeducation Bibliotherapy Stress-coaching Mindfulness-based stress reduction Monitoring and re-assessment
  Vocational rehabilitation is inspired by Individual Placement and Support and is a workplace-oriented intervention with problem-solving conversations as a core element
  Arms: IBBIS integrated MCH and VR

SUMMARY:
The purpose of this study is to investigate the efficacy of 1) a stepped mental health care (MHC) intervention and 2) an integrated mental health care and vocational rehabilitation (VR) intervention for people on sick leave because of burnout, adjustment disorder and psychological stress in Denmark

DETAILED DESCRIPTION:
Background:

Stress disorders have negative effects on workability and have negative effects on both the individual and society. Psychological stress and burnout is not recognized as psychiatric diagnoses, and thus, the estimated prevalence in healthy and sick-listed people is somewhat insecure in Denmark. Together with other common mental disorders, burnout, adjustment disorder and psychological stress are causes of up 40 % of the sick leave claims in Denmark. There is no clear evidence that mental health care alone will provide sufficient support for vocational recovery for this target group. Integrated vocational and health care services have shown good effects on return to work in other Scandinavian countries.

Objective:

The purpose of the Danish IBBIS study is to investigate the efficacy of 1) a stepped mental health care intervention and 2) an integrated mental health care and vocational rehabilitation intervention for people on sick leave because of burnout, adjustment disorder and psychological stress in Denmark.

Method:

This three-arm, randomized, controlled trial is set up to investigate the effectiveness of the stepped mental health care model and the integrated mental health care and vocational rehabilitation intervention for people on sick leave because of burnout, adjustment disorder and psychological stress in Denmark. 603 patients are recruited from Danish job centers in four municipalities. The primary outcome is return to work at 12 months.

Results/discussion:

This study will contribute with new knowledge on vocational recovery and integrated vocational and health care interventions in a Scandinavian context.

ELIGIBILITY:
Inclusion Criteria:

* Burnout OR adjustment disorder OR psychological stress according to 4DSQ
* On sick leave from work or unemployment and have received sick leave benefit for minimum four weeks OR have started a sick leave benefit case which is estimated to last for minimum eight weeks
* Citizen in one of the following municipalities: Copenhagen City, Gladsaxe Municipality, Lyngby-Taarbæk Municipality or Gentofte Municipality
* Danish-speaking
* Given informed consent

Exclusion Criteria:

* Pregnant
* High degree of suicidal ideation
* Dementia
* Alcohol or substance misuse that hinders the person participating in treatment
* Wish to start or continue psychological therapy
* Need for psychiatric treatment in the secondary psychiatric care system
* Medically unstable to a degree that the patient cannot adhere to treatment
* Participant in the research project Collabri
* Attending stress courses in the stress clinics of Copenhagen City
* Assessed by Jobcentre case managers to be dangerous

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 631 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Time to return to work | 12 months
  Time from baseline to first return to work for more than four consecutive weeks

SECONDARY OUTCOMES:
Work | 12 months
  Competitive work 12 months after baseline (yes/no)
Time to return to work | 24 months
  Time from baseline to first return to work for more than four consecutive weeks
Recurrent Sickness Absence | 24 months
  Time from baseline to recurrent sickness absence for more than 8 weeks
Degree of depressive symptoms | 6 months
  Self-assessed anxiety symptoms by the Beck Anxiety Inventory (BDI)
Degree of anxiety symptoms | 6 months
  Self-assessed anxiety symptoms by the Beck Anxiety Inventory (BAI)
Degree of psychological stress symptoms | 6 months
  Self-assessed psychological stress by the Cohen perceived stress scale (PSS)
Work and social functioning | 6 months
  Work and social functioning by the Work and Social Adjustment Scale (WSAS)

OTHER OUTCOMES:
Symptom level | 6, 12 and 24 months
  Symptom level on de four dimensions: Distress, Depression, Anxiety and Somatization by 4-dimensional symptom questionnaire (4DSQ)
Death | 6, 12 and 24 months
  Death and cause of death by register data
Suicidal ideation | 6, 12 and 24 months
  Suicidal ideation by BDI
Life-threatening conditions | 6, 12 and 24 months
  Life-threatening conditions by register data

CONTACTS AND LOCATIONS:
Locations (1):
- Mental Health Services of the Capital Region of Denmark, Copenhagen, Capital Region of Denmark, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hoff A, Poulsen RM, Fisker JP, Hjorthoj C, Nordentoft M, Bojesen AB, Eplov LF. Integrated mental healthcare and vocational rehabilitation for people on sick leave with stress-related disorders: 24-month follow-up of the randomized IBBIS trial. Scand J Work Environ Health. 2023 May 1;49(4):303-308. doi: 10.5271/sjweh.4084. Epub 2023 Mar 5. PMID 36871310
- [Derived] Poulsen R, Fisker J, Hoff A, Hjorthoj C, Eplov LF. Integrated mental health care and vocational rehabilitation to improve return to work rates for people on sick leave because of exhaustion disorder, adjustment disorder, and distress (the Danish IBBIS trial): study protocol for a randomized controlled trial. Trials. 2017 Dec 2;18(1):579. doi: 10.1186/s13063-017-2273-0. PMID 29197404

DOCUMENTS (2):
  • Study Protocol (2019-07-05): https://cdn.clinicaltrials.gov/large-docs/19/NCT02885519/Prot_001.pdf
  • Statistical Analysis Plan (2020-11-30): https://cdn.clinicaltrials.gov/large-docs/19/NCT02885519/SAP_002.pdf